CLINICAL TRIAL: NCT04821609
Title: "Effect of Supervised Resistance Training on Arm Volume and Quality of Life amONG Women at High Risk for Breast Cancer-related Lymphedema: a Study Protocol for a Randomized Controlled Trial (STRONG-B)"
Brief Title: Supervised Resistance TRaining amONG Women at Risk of Breast Cancer Related Lymphedema
Acronym: STRONG-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Universidad de Granada (Other); National Fund for Research and Development in Health, Chile (Other); Hospital Dr Sotero del Rio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA20I0060
Record Dates: First submitted 2021-03-11; First posted 2021-03-29 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Physical Activity; Lymphedema of Upper Arm
Keywords: Resistance training; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training group (Experimental): Twice a week sessions supervised and group, during 12 weeks
  Interventions: Behavioral: Resistance Training
- Control Group (No Intervention): The control group will follow the usual physical therapy management, which does not include resistance training

INTERVENTIONS:
Behavioral: Resistance Training — The resistance training will be for arms and legs, self-loading type, and external weights.
  Arms: Resistance training group

SUMMARY:
Breast cancer (BC) is the most common neoplasm in Chile, and its medical treatment leads to high survival. One-third of survivors will develop BC-related lymphedema. Lymphedema is a chronic condition characterized by increased volume in the ipsilateral arm to surgery. A higher volume is associated with decreased physical functionality and quality of life. Recent studies suggest that resistance training could control arm volume through increased muscle mass development, improving physical functionality and quality of life for patients. To our knowledge, there is no study that has analyzed the effect of a resistance training program among women at risk of BC-related lymphedema on arm volume and quality of life. The purpose of this study is to determine the effect of resistance training on the arm volume and quality of life among women with adjuvant chemotherapy and high risk of BC-related lymphedema compared to a control group with regular physical therapy management, which does not include resistance training.

This is a randomized controlled study. It will be held at the Complejo Asistencial Dr. Sotero del Río, which receives all patients from the South East Metropolitan Health Service. Participants: 106 women receiving adjuvant chemotherapy for BC who have undergone axillary lymph node dissection or with obesity will be recruited. The difference in volume between the arms will be evaluated with optoelectric equipment. Quality of life with The European Organization for Research and Treatment in Cancer Quality of Life C-30 (EORTC QLQ-C30) and the European Organization for Research and Treatment of Breast Cancer-Specific Quality of Life Questionnaire BR23 (EORTC QLQ-BR23) questionnaires, both validated in Chile; the handgrip with a dynamometer; and physical functionality with the six-minute walk test. Volunteers will be randomly assigned to the resistance training group or control group. The resistance training group will consist of twice a week supervised sessions, for 12 weeks. The exercises will be for arms and legs, self-loading type, and with external weights. The control group will follow the usual physical therapy management, which does not include resistance training. Subsequently, volunteers will be evaluated at the third and sixth months after completion of the 12 weeks resistance training program.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with stage I-III breast cancer, histologically confirmed.
* Patients scheduled to receive adjuvant post-operative chemotherapy.
* Partial or total mastectomy with axillary node dissection.
* Partial or total mastectomy with sentinel node dissection with body mass index between 30.0 and 39.9 kg/m2.
* Approval of their treating physician to participate in sub-maximal physiological fitness testing and a low to moderate progressive resistance exercise program.

Exclusion Criteria:

* Inter-limb volume difference greater than 200 ml or 10%.
* Previous antineoplastic treatment (chemotherapy, radiotherapy, or endocrine therapy).
* Breast cancer stage IV
* Unable to participate in an exercise program related to other medical problems.
* Be identified as vigorous exercise behavior related to American College of Sports Medicine recommendations.
* Body mass index lower than 18.5 kg/m2 or greater than 40 kg/m2.
* Pregnancy.
* Fluency and understanding of the Spanish language.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Arms lymphedema Volume on the Perometer System at 3, 6 and 9 months. | Baseline, 3, 6 and 9 months.
  Perometer is considered the gold standard for determining lymphedema volume in research. Is a valid and reliable tool in volume measurement. It determines volume values expressed in milliliters and percentage. A value of 200 mL or 10% difference between one arm and the other is considered significant.
Change from Baseline in Health-related quality of life on questionnaire: The European Organization for Research and Treatment in Cancer (EORTC) Quality of Life C-30 (QLQ-C30) and breast cancer-specific module QLQ-BR23 at 3, 6, and 9 months. | Baseline, 3, 6 and 9 months.
  The QLQ C-30 and specific module QLQ-BR23 are self-administered and validated questionnaires to assess health-related quality of life in patients with breast cancer. Both had been validated in Spanish language and on Chilean population. QLQ-C30 comprises 30 items to assess physical, role, emotional, cognitive, and social functioning. The QLQ-BR23 is a breast-specific module that comprises 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects. All scores were linearly transformed to a 0 to 100 scale. A high functional score represents a high or healthy level of functioning. A high QOL is defined by a high score for global health status or QOL. High symptom scores or items represent more severe symptoms or problems.

SECONDARY OUTCOMES:
Change from Baseline in Hand grip strength on Hydraulic Hand Dynamometer at 3, 6 and 9 months. | Baseline, 3, 6, and 9 months.
  Dynamometer assess the maximal voluntary grip strength (measured in kilograms). Each subject will perform six trials, three in each arm, with an alternating bilateral sequence. The results will be based on the best punctuation of the three trials, respectively. There are normative values in percentiles for healthy Chilean women.
Change from Baseline in Physical Fitness Six minute walk test at 3, 6 and 9 months. | Baseline and 3, 6 and 9 months.
  Six minute walk test is a functional test of sub-maximum cardiorespiratory capacity. Valid and reliable in adults with cancer. Result are expressed in meters. A change of 20-30 meters is considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero, Ph.D, Study Director — Universidad de Granada; Karol Ramírez, Ph.D (c), Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Karol Ramírez, Puente Alto, CO, Chile

REFERENCES:
- [Derived] Ramirez-Parada K, Sanchez C, Cantarero-Villanueva I, Reyes A, Pinto MP, Bravo ML, Montt-Blanchard D, Acevedo F, Walbaum B, Alfaro-Barra M, Barra-Navarro M, Munoz-Flores S, Pinto C, Muniz S, Contreras-Briceno F, Merino T, Merino G. Randomized Trial Assessing Prospective Surveillance and Exercise for Preventing Breast Cancer-Related Lymphedema in High-Risk Patients. Arch Phys Med Rehabil. 2025 Aug;106(8):1163-1172. doi: 10.1016/j.apmr.2025.03.002. Epub 2025 Mar 11. PMID 40081785
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Ramirez-Parada K, Lopez-Garzon M, Sanchez-Rojel C, Petric-Guajardo M, Alfaro-Barra M, Fernandez-Verdejo R, Reyes-Ponce A, Merino-Pereira G, Cantarero-Villanueva I. Effect of Supervised Resistance Training on Arm Volume, Quality of Life and Physical Perfomance Among Women at High Risk for Breast Cancer-Related Lymphedema: A Study Protocol for a Randomized Controlled Trial (STRONG-B). Front Oncol. 2022 Mar 1;12:850564. doi: 10.3389/fonc.2022.850564. eCollection 2022. PMID 35299753